CLINICAL TRIAL: NCT02678364
Title: A Dietary Intervention Study Examining the Effect of Consumption of Vitamin D-enhanced Eggs on Winter-time Vitamin D Status in Adults
Brief Title: Effect of Vitamin D-biofortified Eggs on Wintertime Serum 25-hydroxyvitamin D in Adults: Randomized Controlled Trial
Acronym: EnhanceDeggs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Kevin D. Cashman, Professor of Food and Health, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ECM 4 (y) 07/10/14
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D-biofortified eggs; Vitamin D status; RCT
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control egg group (Placebo Comparator): Two or less control (non-biofortified) eggs per week
  Interventions: Dietary Supplement: Control eggs
- Vitamin D3-eggs group (Active Comparator): Seven vitamin D3-biofortified eggs per week
  Interventions: Dietary Supplement: Vitamin D3 eggs
- 25-Hydroxyvitamin D-eggs group (Active Comparator): 7 25-hydroxyvitamin D-biofortified eggs per week
  Interventions: Dietary Supplement: 25-Hydroxyvitamin D3 eggs

INTERVENTIONS:
Dietary Supplement: Control eggs — Control eggs containing no additional vitamin D beyond norm
  Arms: Control egg group
Dietary Supplement: Vitamin D3 eggs — Vitamin D3-biofortified eggs
  Arms: Vitamin D3-eggs group
Dietary Supplement: 25-Hydroxyvitamin D3 eggs — 25-Hydroxyvitamin D3-biofortified eggs
  Arms: 25-Hydroxyvitamin D-eggs group

SUMMARY:
While there have been a considerable number of studies on the impact of additional vitamin D in the diets of hens on the resulting egg vitamin D content, the effect of consumption of such vitamin D-enhanced eggs on vitamin D status of healthy human subjects has not been tested in a RCT.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effect of consumption of vitamin D3 versus 25-hydroxyvitamin D3 biofortified eggs on winter serum 25(OH)D in adults using a 8-wk randomized controlled trial. This research will provide new data on the potential of vitamin D enriched eggs as a food-based strategy for prevention of vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:

- consenting white men and women aged 45-70 years

Exclusion Criteria:

* consumption of vitamin D-containing supplements throughout the study. planning to take a winter vacation (during the course of the 8-wk intervention) - to a location at which either the altitude or the latitude would be predicted to result in significant cutaneous vitamin D synthesis from solar radiation
* planning to use tanning facilities of any type.
* a severe medical illness,
* allergy to egg products,
* medically advised to limit egg intake in relation to managing hypercholesterolemia,
* hypercalcaemia,
* known intestinal malabsorption syndrome,
* excessive alcohol use,
* the use of medications known to interfere with vitamin D metabolism

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Response of serum total 25-hydroxyvitamin D concentration over 8 weeks of winter | up to 8 weeks

SECONDARY OUTCOMES:
Serum parathyroid hormone | 0 weeks and 8 weeks

OTHER OUTCOMES:
Serum total calcium | 0 weeks and 8 weeks
Serum total cholesterol | 0 weeks and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Cashman, BSc, PhD, Principal Investigator — University College Cork
Locations (1):
- Human Dietary Studies Facility, School of Food and Nutritional Sciences, University College Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hayes A, Duffy S, O'Grady M, Jakobsen J, Galvin K, Teahan-Dillon J, Kerry J, Kelly A, O'Doherty J, Higgins S, Seamans KM, Cashman KD. Vitamin D-enhanced eggs are protective of wintertime serum 25-hydroxyvitamin D in a randomized controlled trial of adults. Am J Clin Nutr. 2016 Sep;104(3):629-37. doi: 10.3945/ajcn.116.132530. Epub 2016 Aug 3. PMID 27488236